CLINICAL TRIAL: NCT01991067
Title: Characterization of Humoral and Cellular Immunity for Tick-borne Encephalitis (TBE) Vaccination in Allogeneic Blood and Marrow Graft Recipients: a Pilot Study
Brief Title: Humoral and Cellular Immunity for TBE Vaccination in Allogeneic HSCT Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Christina Forstner, MD, Associate Professor, PD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EudraCT_2011-002928-41
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Tick Borne Encephalitis
Keywords: Marrow transplant recipients
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — FSME-IMMUN vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HSCT patients / TBE virus vaccine (Active Comparator): Study population: patients who had undergone an allogeneic HSCT 11 to 13 months ago Eligible patients will receive at least two TBE vaccinations (study visit 1 - day 0, study visit 2 -1month after the first vaccination) with a total of two doses of the TBE vaccine FSME-IMMUN®. Whenever possible, the patients will receive complete primary vaccination with a third dose of TBE vaccine (study visit 9 - 9 to 12 months after the first vaccination).
  Interventions: Biological: TBE virus vaccine
- healthy volunteers / TBE virus vaccine (Active Comparator): Clinical healthy volunteers will receive at least two TBE vaccinations (study visit 1 - day 0, study visit 2 -1month after the first vaccination) with a total of two doses of the TBE vaccine FSME IMMUN®. Whenever possible, the volunteers will receive complete primary vaccination with a third dose of TBE vaccine FSME IMMUN® (study visit 9 - 12 months after the first vaccination).
  Interventions: Biological: TBE virus vaccine

INTERVENTIONS:
Biological: TBE virus vaccine — TBE virus vaccine FSME Immun is used in both arms for the study population and the control group
  Other Names: FSME Immun

SUMMARY:
Patients undergoing allogeneic blood and marrow transplantation (HSCT) experience a prolonged period of dysfunctional immunity. Systematic reimmunization is necessary at appropriate time intervals following transplantation to re-establish immunity. Vaccination practices after HSCT remain varied and data sparse. Tick-borne encephalitis (TBE) is one of the most severe infections of the central nervous system caused by a tick-borne flavivirus. There is no specific treatment, and prevention with the vaccine is the only intervention available. To assess the efficacy of TBE vaccination in adult allogeneic HSCT recipients compared to an age-matched and sex-matched control group of healthy volunteers without previous TBE vaccination, a prospective open-label phase II pilot study on humoral and cellular immune responses after use of TBE vaccine (FSME Immun) will be performed. As primary end point the outcome of the neutralization test (NT) against TBE will be assessed in a total of 26 HSCT patients one year after HSCT and in 26 healthy volunteers, namely four weeks after the second vaccination. Therefore, the number of subjects with NT titres against TBE virus >10, assumed to be the threshold for antibody-mediated protection will be evaluated. As secondary endpoints, antibody concentrations of TBE enzyme-linked immunosorbent assay before and four weeks after the second and third vaccination and antibody concentrations of NT against TBE four weeks after primary immunization. To evaluate cellular immune responses, lymphocyte proliferations assays and cytokine detection assays will be performed. In a subgroup analysis, these secondary endpoints will be compared between healthy volunteers, HSCT patients without immunosuppressive treatment and HSCT patients receiving immunosuppressive agents. Additionally, immune reconstitution by analysis of peripheral blood lymphocyte subsets and serum immunoglobulin levels will be evaluated prior to vaccination, after twelve weeks and prior to the third vaccination in HSCT patients only.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects will be eligible for participation in this study if they:

  * Are ≥18 years on the day of screening
  * Had undergone an allogeneic HSCT 11 to 13 months ago (study population)
  * Are clinical healthy without previous TBE vaccination (control group)
  * Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
  * If female and capable of bearing children - have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Subjects will be excluded from participation in this study if they:

  * Have received a TBE vaccination following HSCT
  * Suffer from extremely severe acute graft-versus host disease and therefore receive prednisone >0.5 mg/kg bodyweight as part of a combination therapy or a three agent immunosuppressive treatment (because in these HSCT patients any type of vaccination has to be postponed until immunosuppression is reduced to a double combination or prednisone <0.5 mg/kg bodyweight)
  * Suffer from or have a history of previous TBE virus infection or vaccination, previous dengue virus infection or vaccination against yellow fever or Japanese encephalitis
  * Have any acute febrile illness in the 2 weeks prior to or at the time of enrolment
  * Have a history of severe allergic reactions or anaphylaxis after vaccination
  * If female, are pregnant or lactating.
  * If belonging to the healthy control group, are immunosuppressed (suffer from or have a history of immune mediated diseases, long-term use of corticosteroids, hemodialysis, chronic renal insufficiency, liver cirrhosis Child-Pugh class C, hematooncological malignant disease, solid organ transplant, HSCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Forstner, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Medicine I, Division of Infectious Diseases and Tropical Medicine, Vienna, Austria

REFERENCES:
- [Result] Harrison N, Grabmeier-Pfistershammer K, Graf A, Schwarzinger I, Aberle JH, Stiasny K, Greinix H, Rabitsch W, Kalhs P, Ramharter M, Burgmann H, Forstner C. Humoral immune response to tick-borne encephalitis vaccination in allogeneic blood and marrow graft recipients. NPJ Vaccines. 2020 Jul 24;5(1):67. doi: 10.1038/s41541-020-00215-1. eCollection 2020. PMID 32728481
- [Result] Harrison N, Grabmeier-Pfistershammer K, Graf A, Trapin D, Tauber P, Aberle JH, Stiasny K, Schmidt R, Greinix H, Rabitsch W, Ramharter M, Burgmann H, Pickl WF, Bahrs C. Tick-Borne Encephalitis Specific Lymphocyte Response after Allogeneic Hematopoietic Stem Cell Transplantation Predicts Humoral Immunity after Vaccination. Vaccines (Basel). 2021 Aug 15;9(8):908. doi: 10.3390/vaccines9080908. PMID 34452033

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Started | 19 | 15
Completed | 13 | 10
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Continuous [Median (Full Range); unit: years] | 31 [22 to 61] | 30 [21 to 60] | 30.5 [21 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 11 | 9 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 15 | 34
Body mass index [Median (Full Range); unit: kg/m^2] | 26.9 [19.5 to 39.1] | 22.2 [18.5 to 30.3] | 24.2 [18.5 to 39.1]

OUTCOME MEASURES:

1. Primary Outcome: Outcome of the Neutralization Test (Number of Subjects With Antibody Response Measured by Neutralization Assay)
Description: The Primary endpoint of this study was the antibody Response after TBE-vaccination as measured by neutralization assay four weeks after second vaccination. Antibody response was defined as a Composite endpoint by a NT-titer of >=10, and at least a two-fold increase from baseline (or titer above the highest level of measurement
Time Frame: four weeks after the second vaccination
Population: Patients who received two vaccinations were included in the analysis of the primary end point. Two patients were lost to follow-up after one vaccination and therefore not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 15
Participants | 6 | 14
Statistical Analysis 1: Comparison: HSCT Patients / TBE Virus Vaccine vs Healthy Volunteers / TBE Virus Vaccine; The calculation of the sample size was performed using nQuery 6.1. The primary endpoint was the outcome of the NT 4 weeks after the second vaccination. A Fisher exact tes was calculated to analyze the primary hypothesis on the difference in NT-titer response between patients and controls; Test type: Other — Furthermore, a multivariable logistic regression model was applied accounting for group as well as age, body mass index, and gender as possible influence factors; p < 0.001, Fisher Exact — The threshold for statistical significance was a p-value of <0.05

2. Secondary Outcome: Antibody Response as Measured by TBE-ELISA After Second Vaccination
Description: The antibody response after TBE-vaccination four weeks after second vaccination was measured by ELISA defined by a ELISA titer of >=220 Vienna Units and at least a two-fold increase of titer from baseline
Time Frame: comparison between baseline and four weeks after second vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 15
Participants | 9 | 14
Statistical Analysis 1: Comparison: HSCT Patients / TBE Virus Vaccine vs Healthy Volunteers / TBE Virus Vaccine; A Fisher exact test was calculated to analyze antibody response by ELISA between patients and controls. To measure the Agreement between the NT and ELISA response, Cohens Kappa and the corresponding 95% confidence interval were calculated; Test type: Other; p = 0.02, Fisher Exact

3. Secondary Outcome: Change of Antibody Concentration of NT Titer
Description: Geometric mean fold change of NT titer between baseline and four weeks after third vaccination was compared between HSCT patients and healthy controls
Time Frame: between baseline and four weeks after the third vaccination
Population: Patients who received three vaccinations were included in the analysis. Two patients were lost to follow-up after first vaccination and four patients were lost to follow up after second vaccination therefore not included in the analysis. In the group of healthy volunteers 5 patients were lost to follow-up after second vaccination and therefore not included in the analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean fold change
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 13 | 10
Geometric mean fold change | 3.9 [1.3 to 11.9] | 45.2 [17.5 to 117.0]
Statistical Analysis 1: Comparison: HSCT Patients / TBE Virus Vaccine vs Healthy Volunteers / TBE Virus Vaccine; For titer values the geometric mean was calculated and the corresponding two-sided 95% confidence intervals were constructed by back-transfomration of the CI for the mean of the logarithmically transformed results. To investigate the difference in absolute titer values and geometric mean fold changes between time point and Groups, Wilcoxon tests were performed; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Lymphocyte Proliferation as a Measure of Cellular Immune Response in the Study Population Versus the Control Group Prior Vaccination
Description: Baseline data for lymphocyte proliferation was detected by thymidine incorporation assay after stimulation with albumin-free TBE Antigen. Data was standardized based on unstimulated controls of each participant. The stimulation index is given. The stimulation index is the ratio of the number of proliferating lymphocytes with thymidine incorporation in the presence of antigen to that in absence of antigen. A SI value equal or greater to 3.0 represents relevant lymphocyte proliferation, whereas a SI value <3.0 represents no relevant lymphocyte proliferation.
Time Frame: before vaccination
Population: Patients who received two vaccinations were included in the analysis. Two patients were lost to follow-up after vaccination and therefore not included in the analysis. For the group of healthy volunteers the measure of cellular immune response was optional and therefore only determined in 8 of 15 healthy volunteers.
Measure: Median (Full Range); unit: stimulation index
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 8
stimulation index | 4.2 [1.02 to 69.7] | 0.9 [0.61 to 2.37]

5. Secondary Outcome: Fold Induction in IL13 Cytokine Levels Before Vaccination (Baseline) in the Study Population Versus the Control Group
Description: Determination of secreted IL13 cytokine levels iwas performed using the Luminex System at baseline. Data was standardized based on unstimulated controls of each patient. The fold induction in the presence of TBE antigen to that in absence is given.
Time Frame: before vaccination
Population: Patients who received two vaccinations were included in the analysis. Two patients were last of follow-up after one vaccination and therefore were not included in the analysis. For the group of healthy volunteers the measure of cellular immune response was optional and therefore only determined in 8 of 15 healthy volunteers.
Measure: Median (Full Range); unit: fold induction
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 8
fold induction | 1.0 [0.96 to 98.93] | 0.61 [0.57 to 0.84]

6. Secondary Outcome: Lymphocyte Proliferation as a Measure of Cellular Immune Response in The Study Population Versus the Control Group After Second Vaccination
Description: Data for lymphocyte proliferation was detected by thymidine incorporation assay after stimulation with albumin-free TBE antigen 7 days after the second vaccination. Data was standardized based on unstimulated controls of each participant. The stimulation index is given. The stimulation index is the ratio of the number of proliferating lymphocytes with thymidine incorporation in the presence of antigen to that in absence of antigen. A SI value equal or greater to 3.0 represents relevant lymphocyte proliferation, whereas a SI value <3.0 represents no relevant lymphocyte proliferation.
Time Frame: 7 days after second vaccination
Population: as for outcome 4
Measure: Median (Full Range); unit: stimulation index
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 8
stimulation index | 8.4 [0.7 to 76.6] | 8.3 [1.8 to 23.9]

7. Secondary Outcome: Lymphocyte Proliferation as a Measure of Celluar Immune Response in the Study Population Versus the Control Group After Third Vaccination
Description: Data for lymphocyte proliferation was detected by thymidine incorporation assay after stimulation with albumin-free TBE antigen 7 days after the third vaccination. Data was standardized based on unstimulated controls of each participant. The stimulation index is given. The stimulation index is the ratio of the number of proliferating lymphocytes with thymidine incorporation in the presence of antigen to that in absence of antigen. A SI value equal or greater to 3.0 represents relevant lymphocyte proliferation, whereas a SI value <3.0 represents no relevant lymphocyte proliferation.
Time Frame: 7 days after Third Vaccination
Population: Patients who received three vaccinations were included in the analysis. Two patients were lost to follow-up after first vaccination and four patients were lost to follow up after second vaccination therefore not included in the analysis. For the group of healthy volunteers the measure of cellular immune response was optional and therefore only determined in 5 of 15 healthy volunteers. In the group of healthy volunteers 5 patients were lost to follow-up after second vaccination.
Measure: Median (Full Range); unit: stimulation index
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 13 | 5
stimulation index | 21.0 [0.8 to 109.3] | 13.0 [1.8 to 27.8]

8. Secondary Outcome: Fold Induction in IL13 Cytokine Levels in the Study Population Versus the Control Group After Second Vaccination
Description: Determination of secreted IL13 cytokine levels was performed using the Luminex System 7 days after second vaccination. Data was standardized based on unstimulated controls of each patient. The fold induction in the presence of TBE antigen to that in absence is given.
Time Frame: 7 days after second vaccination
Population: as for outcome 5
Measure: Median (Full Range); unit: fold induction
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 17 | 8
fold induction | 5.6 [1.0 to 180.5] | 2.1 [0.6 to 5.9]

9. Secondary Outcome: Fold Induction in IL13 Cytokine Levels in the Study Population Versus the Control Group After Third Vaccination
Description: Determination of secreted IL13 cytokine levels was performed using the Luminex System 7 days after third vaccination. Data was standardized based on unstimulated controls of each patient. The fold induction in the presence of TBE antigen to that in absence is given.
Time Frame: 7 days after third vaccination
Population: Patients who received three vaccinations were included in the analysis. Two patients were lost to follow-up after first vaccination and four patients were lost to follow-up after second vaccination therefore not included in the analysis. For the group of healthy volunteers the measure of cellular immune response was optional and therefore only determined in 5 of 15 healthy volunteers. In the group of healthy volunteers 5 patients were lost to follow-up after second vaccination.
Measure: Median (Full Range); unit: fold induction
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
Number analyzed (Participants) | 13 | 5
fold induction | 32.3 [0.5 to 153.8] | 3.4 [0.6 to 7.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the whole study period from enrollment to four weeks after third vaccination (Day 298-393 corresponds to 4 weeks after third vaccination)
Arm/Group | HSCT Patients / TBE Virus Vaccine | Healthy Volunteers / TBE Virus Vaccine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 4/19 | 0/15
Other Adverse Events (participants affected / at risk) | 15/19 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSCT Patients / TBE Virus Vaccine (N=19) | Healthy Volunteers / TBE Virus Vaccine (N=15)
cholecystolithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
haemometra (Reproductive system and breast disorders) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 1 (1) | 0 (0)
acute myeloid leukemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSCT Patients / TBE Virus Vaccine (N=19) | Healthy Volunteers / TBE Virus Vaccine (N=15)
local pressure pain (Skin and subcutaneous tissue disorders) | 9 (13) | 5 (7)
local swelling (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
local redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
local induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
shivering (General disorders) | 2 (2) | 1 (1)
fatigue (General disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 3 (4) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
sweating (General disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
cold-like symptoms (General disorders) | 2 (2) | 0 (0)
fever blister (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
increase of Graft-versus-host-disease (skin exanthema) (Immune system disorders) | 1 (1) | 0 (0)
increase of Graft-versus-host-disease (mucosal lesions) (Immune system disorders) | 1 (1) | 0 (0)
subjective tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
skin exanthema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
swelling of parotid gland (Endocrine disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of this study might be the definition of response to vaccination. As the majority of HSCT patients had pre-existing antibodies, the concept of seroconversion was not applicable. Instead, a 2-fold rise in NT titer was used as outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT01991067/Prot_SAP_000.pdf